CLINICAL TRIAL: NCT04637204
Title: Treatment Patterns and Outcomes Among Advanced Renal Cell Carcinoma (aRCC) Patients Treated With Cabozantinib or Axitinib Therapy: Non Interventional, Retrospective Study Using Data From Public Health England's Cancer Analysis System
Brief Title: Real-world Treatment Patterns and Outcomes Among aRCC Patients on Cabozantinib or Axitinib in England
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60000-450
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (4):
- Subgroup 1: Patients with index treatment: cabozantinib treatment post vascular endothelial growth factor (VEGF)-targeted therapy in any line, except axitinib.
  Interventions: Drug: Cabozantinib
- Subgroup 2: Patients with index treatment: axitinib treatment post VEGF-targeted therapy in any line, except cabozantinib.
  Interventions: Drug: Axitinib
- Subgroup 3: Patients with index treatment: cabozantinib treatment post axitinib by line of therapy (2L, 3L, 3L+)
  Interventions: Drug: Cabozantinib
- Subgroup 4: Patients with index treatment: axitinib treatment post cabozantinib by line of therapy (2L, 3L, 3L+)
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Cabozantinib — oral therapy
  Groups: Subgroup 1; Subgroup 3
Drug: Axitinib — oral therapy
  Groups: Subgroup 2; Subgroup 4

SUMMARY:
The present study will aim to describe and understand, in the real-world, the clinical characteristics, treatment patterns and outcomes of advanced renal cell carcinoma (aRCC) patients treated with cabozantinib or axitinib monotherapy in England using the existing data source, Cancer Analysis System (CAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial renal cancer diagnosis
* Patients diagnosed at Stage III or Stage IV (as defined in CAS): as evidence for advanced/metastatic RCC
* For patients with Stage I/II or patients with missing information on Staging
* Patients who received SACT1 treatment following initial renal cancer diagnosis through end of enrolment (31 July 2019)
* Patients who received cabozantinib or axitinib treatment

Exclusion Criteria:

* Diagnosis of concomitant tumour apart from non-melanoma skin cancer in the three years prior to the diagnosis of aRCC
* Less than 18 years of age at the time of initial aRCC diagnosis
* SACT treatment more than 30 days prior to initial aRCC diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult patients diagnosed with aRCC during the study period and identified in the study data source (CAS).
  The study population will comprise two types of aRCC patients:
  * Patients who had advanced disease (Stage III/IV) at diagnosis, and
  * Patients who had non-advanced disease (Stage I/II or missing information on Staging) at diagnosis but advanced at a later date during the study period (proxied by receipt of a SACT treatment indicative of advanced RCC)
Sampling Method: Non-Probability Sample
Enrollment: 1540 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Duration of therapy for the index treatments of interest stratified by line of therapy (LoT) | From start of index treatment up to the end of treatment or start of subsequent therapy during data collection period (01 January 2011 and 31 January 2020)
  Duration of therapy will be measured from the initiation of the index treatment until the projected end date of the index treatment (or start of the subsequent therapy). (subgroups 1 to 4)
Time between subsequent treatment lines | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time gap between the projected end date of the index treatment (cabozantinib or axitinib) until the start of the subsequent treatment. (subgroups 1 to 4)
Sequencing of treatments (any treatments received from aRCC diagnosis until the end of follow up or death) | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Treatment sequencing will be presented using a Sankey diagram that visualises the regimens received within each line of therapy and the number and percentage of patients who received those particular regimens.

SECONDARY OUTCOMES:
Time from aRCC diagnosis to initial SACT initiation | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Defined as the time from diagnosis of aRCC until the start date of the first cycle of the SACT regimen (i.e., 1st LoT start). (subgroups 1 to 4)
Time from RCC diagnosis to initial SACT initiation | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time from RCC diagnosis to initial SACT initiation will be defined as the time from diagnosis of RCC until the start date of the first cycle of the SACT regimen. (subgroups 1 to 4)
Time from RCC diagnosis to treatment initiation of cabozantinib | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time from diagnosis of RCC until the start of the first prescription of cabozantinib. (subgroups 1 and 3)
Time from RCC diagnosis to treatment initiation of axitinib | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time from diagnosis of RCC until the start of the prescription of axitinib.
Time from aRCC diagnosis to treatment initiation of cabozantinib | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time from diagnosis of aRCC until the start of the first prescription of cabozantinib. (subgroups 1 and 3)
Time from aRCC diagnosis to treatment initiation of axitinib | From baseline until the end of data collection period (01 January 2011 and 31 January 2020)
  Time from diagnosis of aRCC until the start of the first prescription of axitinib. (subgroups 2 and 4)
Overall survival (OS) | From start of index treatment until death or end of data collection period (01 January 2011 and 31 January 2020 whichever occurs first
  Time from start of index treatment (cabozantinib/axitinib) until the date of death (from any cause) during the study period. (subgroups 1 to 4)
Landmark survival | 12 months
  Landmark survival will be defined as the time from start of the index treatment until date of death (from any cause) at specific time points (12, 18, and 24 months). (subgroups 1 to 4)
Landmark survival | 18 months
  Landmark survival will be defined as the time from start of the index treatment until date of death (from any cause) at specific time points (12, 18, and 24 months). (subgroups 1 to 4)
Landmark survival | 24 months
  Landmark survival will be defined as the time from start of the index treatment until date of death (from any cause) at specific time points (12, 18, and 24 months). (subgroups 1 to 4)
Time to next treatment (or death) (TTNT) | From start of index treatment until the start of subsequent therapy during data collection period (01 January 2011 and 31 January 2020)
  Time to next treatment (or death) (TTNT) will be defined as the time from start of index treatment until the start of the subsequent LoT (subgroups 1 to 4)
Time to treatment discontinuation (TTTD) | From start of index treatment until discontinuation or death during data collection period (01 January 2011 and 31 January 2020)
  Time to treatment discontinuation (TTTD) will be defined as time from treatment initiation until treatment discontinuation or death. (subgroups 1 to 4)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Facility, Slough, United Kingdom

REFERENCES:
- [Derived] Brown J, Harrow B, Marciniak A, McCarthy C, Houchard A, Cirneanu L, Protheroe A. Cabozantinib and Axitinib After Vascular Endothelial Growth Factor Therapy in Patients with Advanced Renal Cell Carcinoma: A Retrospective Cohort Study from England. Drugs Real World Outcomes. 2024 Jun;11(2):195-207. doi: 10.1007/s40801-023-00415-w. Epub 2024 Jan 24. PMID 38265633